CLINICAL TRIAL: NCT06122168
Title: "Sweet Expectation and Positive Thinking" the Use of the Mandala in the Induction of Labor: a Randomized Clinical Pilot Study.
Brief Title: "Sweet Expectation and Positive Thinking" the Use of the Mandala in the Induction of Labor
Acronym: Mandala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bianca Masturzo (Other)
Responsible Party: Sponsor-Investigator, Bianca Masturzo, Head of Department of Gynaecology and Obstetrics, Ospedale degli Infermi di Biella
Organization: Ospedale degli Infermi di Biella (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CE069/2023
Record Dates: First submitted 2023-10-26; First posted 2023-11-08 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Nulliparity; Induction of Labor Affected Fetus / Newborn
Keywords: nulliparity; mandala; experience; childbirth
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: single center, prospective, randomized trial
Who Masked: Outcomes Assessor
Masking Description: The patients, within the database, will be identified as group A and B; Once the study and the compilation of the database have been completed, this will be delivered to the results evaluation team which will therefore be blinded, not being able to recognize whether group A and B belong to control or intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Standard induction handling plus mandala delivery. The standard management involves, upon admission, a verbal interview with the doctor and midwife regarding the labor induction procedure (Time 1) Time 1 will end with the signing of the consent to participate in the study. Time 2, shortly before the induction, there is a time dedicated to written informed consent relating to the induction, with explanations of possible complications.
  Time 3: once the induction is complete, the patient will be invited to return to the hospital room and where the time for the intervention will start, with the delivery of the mandala and colours. During the phases preceding the start of labour, except for the time dedicated to coloring the mandala, the patient will be subjected to standard care management, as required by the ward induction protocol.
  Interventions: Other: Mandala
- Control Group (Active Comparator): Will follow all the standard management of hospitalization, informed consent and post-induction (time 1, 2 and 3) foreseen for the intervention group, but will not receive the mandala.
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Mandala — verbal interview, standard health care, sheet of paper showing a mandala to be colored at will
  Arms: Intervention Group
Other: Standard care — verbal interview and standard health care
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of an artistic tool, the mandala, in a population of pregnant women (nulliparous) undergoing labor induction.

The main questions it aims to answer are:

* Does using the mandala during labor induction improve the birth experience?
* Does the use of the mandala during the induction of labor improve the outcome of the birth and the demand for analgesia? Participants in the intervention group will receive standard treatment plus coloring mandala, those in the control group only standard treatment.

DETAILED DESCRIPTION:
Labor induction is one of the most frequent gestures in the daily clinical practice of an obstetrics department. In recent decades there has been an increase in this practice, the reasons for which are not entirely understandable, but being a medical intervention it must be as appropriate as possible. The induction of labor is implemented in order to interrupt the evolution of the pregnancy and the goal is to obtain an active labor in conditions of maternal-fetal well-being (SIGO Guidelines 2022). WHO recommends that women's experiential experience with respect to their nursing care be considered of equal importance to clinical care. A positive birth experience is a good indicator for women who decide to have more children and is positively related to the establishment of the mother-infant bond as well as maternal confidence in breastfeeding. Consequently, a negative birth experience in addition to negatively influencing the decision to have another child, also affects the well-being of the mother and leads to high levels of anxiety. A study has shown that the feeling of control and participation in choosing one's birth experience is related to a positive birth experience. From the point of view of the perception of safety and the sense of participation during labour, induced patients appear to have lower levels than women in spontaneous labour, this should sensitize the midwives and health professionals involved in the process, to provide better support.

Study design: randomized clinical pilot study in parallel groups, patients will be assigned to the two groups through the sealed envelope method.

Intervention: Intervention group. Patients assigned to this group will receive standard induction management plus mandala delivery. The standard management provides, upon admission, a verbal interview with the doctor and midwife regarding the labor induction procedure (Time 1), specifically:

* explanation of the diagnosis requiring labor induction;
* induction times;
* induction methods;
* type of assistance and obstetric/medical surveillance;
* possibility of support from the partner;
* information related to the stay in the ward;
* verbal and written information on the study and request for participation. Time 1 will end with the signing of the consent to participate in the study. Time 2, shortly before the induction, there is a time dedicated to written informed consent relating to the induction, with explanations of possible complications. Time 3: once the induction is over, the patient will be invited to return to the hospital room where the time of the intervention will start, with the delivery of the mandala and colours. During the phases preceding the start of labour, except for the time dedicated to coloring the mandala, the patient will be subjected to standard care management, as required by the ward induction protocol. Control group: will follow all the standard management of hospitalization, informed consent and post induction (time 1, 2 and 3) foreseen for the intervention group, but will not receive the mandala.

Sample size estimation: based on literature data which report an average CEQ value of 2.9 in nulliparous women and calculating the variance on the basis of a standard deviation equal to 0.6, with a 95% confidence level and a power of 80%, it is estimated that 49 patients need to be enrolled to observe a difference between CEQ scale scores of 0.34 points.

Allocation: in order to be able to assign the patients to one of the two groups, sealed envelopes will be generated, equal to the number of participants expected in the study. Inside the envelope it will be stated which group the patient will participate in by the wording "CONTROL" or "INTERVENTION", it will not be possible to change the allocation sequence based on the patient's or team's preferences. The sealed envelopes will be created by a team separate from the one that will take care of the data, specifically by the person set out as responsible for the "Conceptualization, methodology, writing and review" part, who will not participate in any way in the clinical management- patient care and care and data management. Once the envelopes have been generated, which will be identical in shape, color and content, so as to make them unrecognizable, they will be mixed, delivered and stored in a locked drawer that can only be opened by the team designated as responsible for data care. After opening the sealed envelope, the allocation to one of the two groups will be established by the doctor who will also establish the need for hospitalisation, diagnose the need for induction and have the consent to participate in the study signed. The sealed envelope will be delivered by the team responsible for data care, only after completing all the procedures foreseen in time 1, and shortly before delivering the patient to the inpatient ward.

Recruitment: recruitment to the study will take place only after verification of the inclusion criteria set out in the following protocol. There will be an initial selection by the obstetrics/gynecological staff, made aware of all the parts of the protocol, who will be able to recognize a patient with the characteristics suitable for participation in the study. The team indicated as "project and investigation administrator" will then be contacted, which will have the final responsibility for including or excluding the patient, after careful evaluation of all the criteria set out.

Delivery of the intervention: once the hospitalization phases, foreseen at time 1 and the recruitment and allocation phases have been completed, the patient will be taken to the hospital ward, in this phase the ward midwives will be informed with respect to the group to which they belong, so that they can the mandala, if it is the intervention group, vice versa the standard management will start. At the end of the hospitalization, the medical records of the patients in the study will be handed over to the team responsible for data care.

Data management A specially created database will be compiled, in which the main characteristics of the enrolled patients will be collected (age, week of gestation, reason for induction, presence of partners, educational qualifications, etc.). Furthermore, the data of the answers to the anonymous questionnaire and those relating to the secondary outcomes will be collected, through the patient's medical record, which will be kept separately, in a locked drawer, by the team responsible for data care. The team designated for "formal, methodological and data management analysis" will take care of compiling the database. The patients, within the database, will be identified as group A and B; Once the study and the compilation of the database have been completed, this will be delivered to the results evaluation team which will therefore be blinded, not being able to recognize whether group A and B belong to control or intervention.

Blindness

* Allocation: will take place blindly as specified in the previous paragraph;
* Study participants: they will not be blinded, since the administration of the mandala cannot be hidden;
* Assistance providers: they will not be blinded for the above reason;
* Outcome evaluators and data analysis: blinded thanks to data entry with group A and B methods and not as a control and intervention.

Statistical analysis plan: possible confounding variables will be collected in a questionnaire at baseline, and, in the case of statistically significant differences between the experimental and control group, an adjustment will be made by stratification or logistic regression.

Primary outcome: the difference between the mean of the CEQ scores in the two groups and the relative standard deviation will be estimated, in order to obtain an evidence-based measure based on the difference between means weighted by the sample size with the relative 95% confidence intervals (weighted mean difference - WMD); the estimate will be made both for the overall score and for the specific area.

Secondary outcomes: the results will be presented as cumulative incidences in the two groups and relative risks with the relative 95% confidence intervals for the dichotomous variables; for the continuous variables, means will be presented with the relative standard deviations in the two groups and the WMD with relative 95% confidence interval will be used as a summary measure.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* hospitalized for the need to induce labor for medical reasons
* single fetus in cephalic presentation
* gestational age ≥ 37 weeks
* having provided written consent to participate in the study

Exclusion Criteria:

* inductions requiring the initial use of oxytocin
* prenatal fetal complications such as severe intrauterine growth restriction (IUGR)
* suspicious or non-reassuring cardiotocography upon entry to the ward
* inability to understand the questionnaire and the information material provided
* all hospitalizations for primary causes other than induction

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2025-02-16 (Actual); Study Completion 2025-02-16 (Actual)

PRIMARY OUTCOMES:
Experience of childbirth through the Childbirth experience questionnaire (CEQ) | 24 hours after giving birth
  Evaluate whether the use of the mandala affects the woman's experience with birth through a questionnaire consisting of 22 questions, the Childbirth experience questionnaire (CEQ). The rating range is 1 to 4 with higher ratings reflecting more positive experiences.

SECONDARY OUTCOMES:
Evaluate the outcome of the birth through the patient's medical records, specifically whether it ended in spontaneous birth or cesarean section or instrumental birth. | up to 24 weeks
  At the end of the patient's hospital stay, subjected to the study, the given outcome of the birth will be retrieved from the patient's medical record, where the type of birth is already usually described: spontaneous or cesarean section or instrumental. The data will be inserted into a specially created database.
Use and request by the patient in the study of epidural analgesia during labor | up to 24 weeks
  At the end of the patient's hospitalization, the request and use of epidural analgesia during childbirth will be noted in the patient's medical record, where they are normally reported. The data will be entered into a specially created database.

CONTACTS AND LOCATIONS:
Overall Officials: bianca masturzo, Md, PhD, Principal Investigator — Ospedale degli Infermi di Biella
Locations (1):
- Bianca Masturzo Ospedale degli Infermi, Ponderano, Biella, Italy

IPD SHARING:
Plan to Share IPD: Yes
The data will be made available through a database, created to collect data during all phases of the study.
Supporting Information: Study Protocol, CSR
Time Frame: At the end of the study
Access Criteria: Participants centers and to other researchers who will ask the managers for details of the study data
URL: https://aslbi.piemonte.it/reparti-e-servizi/informazioni-generali-sui-servizi/ostetricia-e-ginecologia/

REFERENCES:
- [Background] Tuncalp Ӧ, Were WM, MacLennan C, Oladapo OT, Gulmezoglu AM, Bahl R, Daelmans B, Mathai M, Say L, Kristensen F, Temmerman M, Bustreo F. Quality of care for pregnant women and newborns-the WHO vision. BJOG. 2015 Jul;122(8):1045-9. doi: 10.1111/1471-0528.13451. Epub 2015 May 1. No abstract available. PMID 25929823
- [Background] Mercer RT, Ferketich SL. Maternal-infant attachment of experienced and inexperienced mothers during infancy. Nurs Res. 1994 Nov-Dec;43(6):344-51. PMID 7971298
- [Background] Waldenstrom U, Hildingsson I, Ryding EL. Antenatal fear of childbirth and its association with subsequent caesarean section and experience of childbirth. BJOG. 2006 Jun;113(6):638-46. doi: 10.1111/j.1471-0528.2006.00950.x. PMID 16709206
- [Background] Cook K, Loomis C. The Impact of Choice and Control on Women's Childbirth Experiences. J Perinat Educ. 2012 Summer;21(3):158-68. doi: 10.1891/1058-1243.21.3.158. PMID 23730127
- [Background] Coates R. Attitudes of pregnant women and healthcare professionals to labour induction and obtaining consent for labour induction. Best Pract Res Clin Obstet Gynaecol. 2021 Nov;77:64-75. doi: 10.1016/j.bpobgyn.2021.08.008. Epub 2021 Aug 27. PMID 34625350
- [Background] Coates D, Goodfellow A, Sinclair L. Induction of labour: Experiences of care and decision-making of women and clinicians. Women Birth. 2020 Feb;33(1):e1-e14. doi: 10.1016/j.wombi.2019.06.002. Epub 2019 Jun 15. PMID 31208865
- [Background] Dupont C, Blanc-Petitjean P, Cortet M, Gaucher L, Salome M, Carbonne B, Ray CL. Dissatisfaction of women with induction of labour according to parity: Results of a population-based cohort study. Midwifery. 2020 May;84:102663. doi: 10.1016/j.midw.2020.102663. Epub 2020 Feb 14. PMID 32092607
- [Background] Schwarz C, Gross MM, Heusser P, Berger B. Women's perceptions of induction of labour outcomes: Results of an online-survey in Germany. Midwifery. 2016 Apr;35:3-10. doi: 10.1016/j.midw.2016.02.002. Epub 2016 Feb 8. PMID 27060393
- [Background] Place K, Kruit H, Rahkonen L. Comparison of primiparous women's childbirth experience in labor induction with cervical ripening by balloon catheter or oral misoprostol - a prospective study using a validated childbirth experience questionnaire (CEQ) and visual analogue scale (VAS). Acta Obstet Gynecol Scand. 2022 Oct;101(10):1153-1162. doi: 10.1111/aogs.14433. Epub 2022 Aug 7. PMID 35933726
- [Background] Evans K, Sands G, Spiby H, Evans C, Pallotti P, Eldridge J. A systematic review of supportive interventions to promote women's comfort and well-being during induction of labour. J Adv Nurs. 2021 May;77(5):2185-2196. doi: 10.1111/jan.14711. Epub 2020 Dec 14. PMID 33314297
- [Background] Adler K, Rahkonen L, Kruit H. Maternal childbirth experience in induced and spontaneous labour measured in a visual analog scale and the factors influencing it; a two-year cohort study. BMC Pregnancy Childbirth. 2020 Jul 21;20(1):415. doi: 10.1186/s12884-020-03106-4. PMID 32693773
- [Background] Joensuu JM, Saarijarvi H, Rouhe H, Gissler M, Ulander VM, Heinonen S, Torkki P, Mikkola TS. Maternal childbirth experience and induction of labour in each mode of delivery: a retrospective seven-year cohort study of 95,051 parturients in Finland. BMC Pregnancy Childbirth. 2022 Jun 23;22(1):508. doi: 10.1186/s12884-022-04830-9. PMID 35739476